CLINICAL TRIAL: NCT03625778
Title: A Randomized, Blinded, Placebo-controlled Study to Assess Pharmacokinetics, Safety, and Tolerability of Ascending Doses of MEDI0382 in Non-diabetic Obese Subjects
Brief Title: A Study to Assess Safety, Tolerability, and Pharmacokinetics of MEDI0382 in Non-diabetic Obese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D5672C00001
Record Dates: First submitted 2018-07-27; First posted 2018-08-10 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Obesity
Keywords: Obesity; MEDI0382; Overweight
MeSH Terms: conditions — Obesity; Overweight | interventions — cotadutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: In Cohort 1 participants are blinded however site staff, investigator, and sponsor are unblinded. In Cohorts 2 and 3 participants, investigators, site staff, and clinical research organization staff are blinded and sponsor is unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Placebo Cohort 1 (Placebo Comparator): Participants will receive subcutaneous (SC) placebo matched to MEDI0382 Cohort 1 once daily for 9 weeks.
  Interventions: Drug: Placebo
- MEDI0382 Cohort 1 (Experimental): Participants will receive SC MEDI0382 titrated doses of Dose 1 to 7 once daily (7-step titration/ 1 week per dose) from Weeks 1 to 7 followed by additional treatment of SC MEDI0382 Dose 7 once daily from Weeks 7 to 9.
  Interventions: Drug: MEDI0382
- Placebo Cohort 2 (Placebo Comparator): Participants will receive SC placebo matched to MEDI0382 Cohort 2 once daily for 14 weeks.
  Interventions: Drug: Placebo
- MEDI0382 Cohort 2 (Experimental): Participants will receive SC MEDI0382 titrated doses of Doses 1, 2, 3, 5, and 7 once daily (5-step titration/ 2 week per dose) from Weeks 1 to 10 followed by additional treatment of SC MEDI0382 Dose 7 once daily from Weeks 11 to 14.
  Interventions: Drug: MEDI0382
- Placebo Cohort 3 (Placebo Comparator): Participants will receive SC placebo matched to MEDI0382 Cohort 3 once daily for 18 weeks.
  Interventions: Drug: Placebo
- MEDI0382 Cohort 3 (Experimental): Participants will receive SC MEDI0382 titrated doses of Doses 1, 8, 4, and 7 once daily (4-step titration/ 4 week per dose) from Weeks 1 to 16 followed by additional treatment of SC MEDI0382 Dose 7 once daily from Weeks 17 to 18.
  Interventions: Drug: MEDI0382

INTERVENTIONS:
Drug: MEDI0382 — MEDI0382 will be administered subcutaneously daily according to the MEDI0382 cohorts.
  Other Names: Cotadutide
  Arms: MEDI0382 Cohort 1; MEDI0382 Cohort 2; MEDI0382 Cohort 3
Drug: Placebo — Placebo will be administered subcutaneously daily according to the Placebo cohorts.
  Arms: Placebo Cohort 1; Placebo Cohort 2; Placebo Cohort 3

SUMMARY:
This is a Phase 1, randomized, blinded, placebo-controlled study in up to approximately 51 non-diabetic obese participants with a body mass index (BMI) ≥ 35 kg/m^2. The participants will be observed among 3 separate cohorts and participate in the study for up to approximately 27 weeks, including a screening period (including a run-in), treatment period, and safety follow-up.

DETAILED DESCRIPTION:
This is a Phase 1, randomized, blinded, placebo-controlled study in up to approximately 51 non-diabetic obese participants with a BMI ≥ 35 kg/m2. Participants will be blinded, but investigators/site staff and sponsor will be unblinded for Cohort 1. In Cohorts 2 and 3 participants, investigators, and contract research organization personnel are blinded to investigational product and sponsor is unblinded. The participants will participate in the study for up to approximately 27 weeks, including a screening period (including a run-in), treatment period, and safety follow-up.

Participants will be randomized 4:1 to MEDI0382 (n=12) or placebo (n=3) for Cohort 1 and randomized 2:1 to MEDI0382 (n=12) or placebo (n=6) for Cohorts 2 and 3. In Cohort 1 participants randomized to MEDI0382 or placebo will be dosed daily with a weekly titration schedule until the highest clinically tolerated dose (CTD) is established. In Cohort 2 participants randomized to MEDI0382 or placebo will be dosed daily with a 2 week titration schedule up to the highest CTD is established in Cohort 1. In Cohort 3 participants randomized to MEDI0382 or placebo will be dosed daily with a 4 week participants schedule up to the highest CTD established in Cohort 1. Once the highest CTD is identified, participants will continue on the highest CTD for an additional 2 weeks of treatment for Cohort 1 and 3 and additional 4 weeks treatment for Cohort 2. All participants will return 28 days post last dose for a safety follow-up visit.

ELIGIBILITY:
Key Inclusion Criteria:

1. Provision of written informed consent
2. Male and female participants age 18 through 65 years
3. BMI ≥ 35 kg/m^2
4. Hemoglobin A1c level of < 6.5%
5. Female participants must have a negative pregnancy test and must not be lactating.
6. Females of childbearing potential using appropriate birth control to avoid pregnancy during the study.
7. Stable body weight
8. Willing and able to adhere to the visit/protocol schedule, including following lifestyle advice with respect to diet and exercise for the duration of the study
9. Willing and able to self-administer daily SC injections following an initial self-injection training

Key Exclusion Criteria:

1. Any clinically important illness, medical/surgical procedure, or trauma within 4 weeks prior to Study Day 1 dosing.
2. Any condition that, in the opinion of the investigator, would interfere with the evaluation of the investigational product or interpretation of participants safety or study results.
3. Active participation in any other investigation clinical study.
4. Any prescription or non-prescription drugs for weight loss including herbal or other dietary supplements used within the past 3 months prior to screening.
5. Previous glucagon-like peptide-1 (GLP-1) use within 3 months prior to screening.
6. Any positive results for serum hepatitis B surface antigen, hepatitis C virus antibody and/or human immunodeficiency virus (HIV) antibody at screening.
7. Laboratory tests results as specified in the protocol (laboratory tests may be repeated once for confirmation of out of range values at screening).
8. Significant hepatic or renal impairment
9. Poorly controlled hypertension
10. Known or suspected history of drug or alcohol abuse within the past year or positive current test
11. Previous surgical procedures for weight loss

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2018-08-14 (Actual); Primary Completion 2019-08-25 (Actual); Study Completion 2019-08-25 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs) for Cohorts 1, 2, and 3 | From Day 1 through 28 days after the last dose of study drug (approximately 13, 18, and 22 weeks for Cohorts 1, 2, and 3, respectively)
  An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. The TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug.
Number of Participants With Abnormal Clinical Laboratory Parameters Reported as TEAEs for Cohorts 1, 2, and 3 | From Day 1 through 28 days after the last dose of study drug (approximately 13, 18, and 22 weeks for Cohorts 1, 2, and 3, respectively)
  Number of participants with abnormal clinical laboratory parameters reported as TEAEs are reported. Abnormal clinical laboratory parameters were defined as any abnormal finding during analysis of hematology, clinical chemistry, and urinalysis.
Number of Participants With Abnormal Vital Signs and Physical Examinations Reported as TEAEs for Cohorts 1, 2, and 3 | From Day 1 through 28 days after the last dose of study drug (approximately 13, 18, and 22 weeks for Cohorts 1, 2, and 3, respectively)
  Number of participants with abnormal vital signs (body temperature, blood pressure, heart rate, and respiratory rate) and physical examinations reported as TEAEs are reported.
Number of Participants With Abnormal Electrocardiogram (ECG) Parameters Reported as TEAEs for Cohorts 1, 2, and 3 | From Day 1 through 28 days after the last dose of study drug (approximately 13, 18, and 22 weeks for Cohorts 1, 2, and 3, respectively)
  Number of participants with abnormal ECG parameters reported as TEAEs are reported.
Change in Blood Pressure from Baseline to End of Dosing as Measured by Telemetry for Cohort 1 | From Baseline (Day -1) through end of dosing (Day 63)
  Telemetry is the process of recording and transmitting the vital readings (temperature, blood pressure, pulse rate, and respiratory rate). It is used to continuously monitor vital reading as a real-time safety measure. Mean change in blood pressure from baseline to end of dosing measured by telemetry for Cohort 1 are reported.
Change in Respiratory Rate from Baseline to End of Dosing as Measured by Telemetry for Cohort 1 | From Baseline (Day -1) through end of dosing (Day 63)
  Telemetry is the process of recording and transmitting the vital readings (temperature, blood pressure, pulse rate, and respiratory rate). It is used to continuously monitor vital reading as a real-time safety measure. Mean change in respiratory rate from baseline to end of dosing measured by telemetry for Cohort 1 are reported.
Change in Pulse Rate from Baseline to End of Dosing as Measured by Telemetry for Cohort 1 | From Baseline (Day -1) through end of dosing (Day 63)
  Telemetry is the process of recording and transmitting the vital readings (temperature, blood pressure, pulse rate, and respiratory rate). It is used to continuously monitor vital reading as a real-time safety measure. Mean change in pulse rate from baseline to end of dosing measured by telemetry for Cohort 1 are reported.
Change in Temperature from Baseline to End of Dosing as Measured by Telemetry for Cohort 1 | From Baseline (Day -1) through end of dosing ( Day 63)
  Telemetry is the process of recording and transmitting the vital readings (temperature, blood pressure, pulse rate, and respiratory rate). It is used to continuously monitor vital reading as a real-time safety measure. Mean change in temperature from baseline to end of dosing measured by telemetry for Cohort 1 are reported.

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of MEDI0382 for Cohort 1 | Predose (-5 minutes) and 1, 2, 4, 6, 8, 12, and 24 hours postdose on Days 7, 14, 21, 28, 35, 42, and 49 for MEDI0382 Doses 1 to 7, respectively
  The Cmax of MEDI0382 (Cotadutide) for MEDI0382 Doses 1 to 7 for Cohort 1 are reported.
Cmax of MEDI0382 Dose 1 on Day 1 for Cohort 1 | Predose (-5 minutes) and 1, 2, 4, 6, 8, 12, and 24 hours postdose on Day 1
  The Cmax of MEDI0382 Dose 1 for Cohort 1 is reported.
Area Under the Concentration-time Curve at the end of the Dosing interval (AUCτ) of MEDI0382 for Cohort 1 | Predose (-5 minutes) and 1, 2, 4, 6, 8, 12, and 24 hours postdose on Days 7, 14, 21, 28, 35, 42, and 49 for MEDI0382 Doses 1 to 7, respectively
  The AUCτ of MEDI0382 for MEDI0382 Doses 1 to 7 for Cohort 1 are reported.
AUCτ of MEDI0382 Dose 1 on Day 1 for Cohort 1 | Predose (-5 minutes) and 1, 2, 4, 6, 8, 12, and 24 hours postdose on Day 1
  The AUCτ of MEDI0382 Dose 1 for Cohort 1 is reported.
Time to Maximum Observed Plasma Concentration (Tmax) of MEDI0382 for Cohort 1 | Predose (-5 minutes) and 1, 2, 4, 6, 8, 12, and 24 hours postdose on Days 7, 14, 21, 28, 35, 42, and 49 for MEDI0382 Doses 1 to 7, respectively
  The Tmax of MEDI0382 for MEDI0382 Doses 1 to 7 for Cohort 1 are reported.
Tmax of MEDI0382 Dose 1 on Day 1 for Cohort 1 | Predose (-5 minutes) and 1, 2, 4, 6, 8, 12, and 24 hours postdose on Day 1
  The Tmax of MEDI0382 Dose 1 for Cohort 1 is reported.
Plasma Concentration of MEDI0382 for Cohorts 2 and 3 | Cohort 2: predose and 6 hours postdose on Days 1, 15, 29, 43, and 57 for MEDI0382 Doses 1, 2, 3, 5, and 7, respectively; Cohort 3: predose and 6 hours postdose on Days 1, 29, 57, and 85 for MEDI0382 Doses 1, 8, 4, and 7, respectively
  Plasma concentration of MEDI0382 for predose and 6 hours postdose for Cohorts 2 and 3 are reported.
Plasma Concentration of MEDI0382 Dose 7 on Day 71 for Cohort 2 and MEDI0382 Dose 7 on Day 113 for Cohort 3 | Cohort 2: predose and 6 hours postdose on Day 71 for MEDI0382 Dose 7; Cohort 3: predose and 6 hours postdose on Day 113 for MEDI0382 Dose 7
  Plasma concentration of MEDI0382 Dose 7 for predose and 6 hours postdose on Day 71 for Cohort 2 and on Day 113 for Cohort 3 are reported.
Number of Participants With Positive Anti-Drug Antibodies (ADA) to MEDI0382 in all Cohorts | Predose on Baseline (Day -1) and follow-up visit (28 days after the last dose) for each cohort; predose on Days 28 and 50 for Cohort 1, on Days 7, 28, 71, 98 for Cohort 2, and on Days 7, 28, 71, 126 for Cohort 3
  Number of participants with positive ADA to MEDI0382 are reported.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Research Site, Daytona Beach, Florida
  - Research Site, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Results of this clinical trial are available on www.astrazenecaclinicaltrials.com — https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Search